PROTOCOL TITLE: Anterior-segment OCT (AS-OCT) and intraoperative OCT (iOCT) for transconjunctival needle revision (TCNR) of trabeculectomy bleb

## PRINCIPAL INVESTIGATOR:

Angelo P. Tanna, MD

**Department of Ophthalmology** 

Northwestern University Feinberg School of Medicine

Telephone Number: 312-908-8152

Email Address: atanna@northwestern.edu

**VERSION DATE: 04/16/2021** 

## **STUDY SUMMARY:**

| Investigational Agent(s) | N/A |
|---|---|
| (Drugs or Devices) | |
| IND / IDE / HDE # | |
| | Children |
| | Children who are wards of the state |
| | Adults Unable to Consent |
| Indicate | Cognitively Impaired Adults |
| Special Population(s) | Neonates of Uncertain Viability |
| | Pregnant Women |
| | Prisoners (or other detained/paroled individuals) |
| | Students/Employees |
| Sample Size | Prospective study: 25 Subjects |
| | Retrospective study (historical controls): 25 subjects |
| Funding Source | Department of Ophthalmology |
| Turiumg Source | Illinois Society for the Prevention of Blindness |
| | ⊠Written |
| Indicate the type of consent | Verbal/Waiver of Documentation of Informed Consent |
| to be obtained | Waiver of HIPAA Authorization |
| | Waiver/Alteration of Consent Process |

Version Date: 04/16/2021  HRP-593 / v03152019

| Site | Lead Site ( For A Multiple Site Research Study) |
|----------------------------|-------------------------------------------------|
| Site | ☐ Data Coordinating Center (DCC) |
| Research Related Radiation | Yes |
| Exposure | ⊠ No |
| DSMB / DMC / IDMC | Yes |
| | □No |

#### **OBJECTIVES:**

The aim of the research is to assess the surgical success, feasibility and utility of pre-operative Anterior Segment Optical Coherence Tomography (AS-OCT) and intraoperative Optical Coherence Tomography (iOCT) in trans-conjunctival needle revision (TCNR) of trabeculectomy bleb. Furthermore, we want to assess whether AS-OCT can be used to identify characteristics of trabeculectomy blebs that are associated with successful surgical outcomes.

To undergo this study, we will conduct a prospective study of patients who consent to AS-OCT and iOCT revision of TCNR. We will compare the outcomes of these patients with retrospectively identified, historical controls (i.e. patients who underwent TCNR by the same surgeon without AS-OCT or iOCT assistance).

We hypothesize that information gained from pre-operative AS-OCT and intraoperative OCT will aid with intraoperative decision-making for TCNR of trabeculectomy bleb and will thereby improve surgical outcomes. We also hypothesize that preoperative AS-OCT can be used to identify features of trabeculectomy bleb that can predict success with iOCT-assisted TCNR. More specifically, we hypothesize that filtering blebs with more extensive scarring as seen on pre-operative AS-OCT will benefit from iOCT.

### **BACKGROUND:**

Trabeculectomy is one of the most commonly performed glaucoma procedures performed to control IOP with approximately 18,000 operations performed in US Medicare beneficiaries

Version Date: 04/16/2021  HRP-593 / v03152019

STU00213080

alone in 2012.¹ One complication of trabeculectomy surgery is the formation of subconjunctival

and episcleral fibrosis, which occurs as part of the wound healing process and can result in

fibrosis of the filtering bleb and failure. Transconjunctival needle revision (TCNR) aims to lyse

subconjunctival adhesions and reestablish adequate aqueous humor flow from the anterior

chamber to the subconjunctival space. One study reported 17% of trabeculectomies require

bleb-needling revision.<sup>2</sup> During TCNR the surgeon is able to visualize the trajectory of the

needle or blade under the conjunctiva; however, detection of the fibrotic tissue and

determination as to whether that tissue has been adequately lysed is difficult, limiting the

success rate of the procedure.

Anterior segment optical coherence tomography (AS-OCT) allows for detailed assessment of the

internal morphology of the bleb. Studies have utilized AS-OCT to assess morphological features

of the bleb and correlate it with surgical success.<sup>3,4,7</sup> A small case series reported the utility of

AS-OCT for pre-operative planning for bleb revision, in particular, identifying safe access sites

and minimizing conjunctival dissection.<sup>5</sup>

More recently, real time OCT integrated with operative microscope has become available.

Intraoperative OCT (iOCT) has been utilized extensively in retinal surgery and corneal surgery.<sup>6</sup>

Dada et al., described performing iOCT-guided TCNR in 2 patients with failed trabeculectomy

blebs without intraoperative or postoperative complications. These authors report they were

able to obtain a detailed view of the bleb wall and assess the depth and location of the needle,

which permitted better lysis of adhesions. A pilot study by Kumar et al., reported one case of

TCNR in which iOCT was used to demonstrate the extent of adhesions and loculations inside the

bleb at the beginning of the procedure, and the lysis of these adhesions and formation of large

single hyporeflective cavity inside the bleb at the end of the procedure.8 These small case

studies suggest a role of iOCT imaging for TCNR, however, further research is needed to assess

its feasibility and utility for routine use.

STUDY ENDPOINTS:

Version Date: 04/16/2021

 HRP-593 / v03152019

STU00213080

Results from the following tests obtained as part of this study:

1. Spectralis Anterior-segment OCT (AS-OCT) (Heidelberg Engineering) available in Lavin 15th

floor Ophthalmology clinic

2. Digital microscope integrated with Intraoperative OCT (Zeiss Artevo 800, Carl Zeiss Meditec

AG) available in the Lavin 11th floor operating room

The primary outcome will be surgical success, defined as a 20% reduction in unmedicated IOP

below the pre-operative baseline at the post-operative visits (POD1, POM1, POM3). The success

rate will be compared to a cohort of historical controls comprised of a consecutive series of

age- and race-matched subjects who underwent TCNR in the operating room by the same

surgeon, with the same intraoperative anti-fibrotic therapy, without AS-OCT or iOCT imaging

during a five-year time period from 6/1/2015 to 6/1/2020.

The secondary outcomes will be feasibility and utility of intraoperative OCT. Feasibility will be

defined as the percentage of cases with successful imaging of the bleb with iOCT. Utility will be

defined as the percentage of cases in which iOCT changed surgical decision-making.

Intraoperative OCT will be used to determine whether adhesions have been completely lysed

and/or whether further lysis of adhesions is necessary. A survey with set of questions based on

prior literature<sup>6</sup> will be used to assess these parameters.

We will also assess whether findings seen with pre-operative AS-OCT can predict what type of

blebs will benefit from iOCT-assisted TNCR. Features of AS-OCT and iOCT imaging that will be

assessed include quality of image capture, visualization of surgical site, and characteristics of

the bleb. Characteristics of the surgical site include bleb height, internal reflectivity, location

and number of adhesions, and presence of cysts, cavities, and fistulas.

STU00213080

STUDY INTERVENTION(S) / INVESTIGATIONAL AGENT(S):

This prospective study will include approximately 25 patients with open-angle glaucoma who

will undergo TCNR of trabeculectomy bleb by a glaucoma specialist at Northwestern Medicine.

These patients will have a history of glaucoma and failed trabeculectomy bleb (as evidenced by

clinical features and elevated IOP). During routine clinic visit, the patient will undergo lit lamp

grading of bleb by Indiana Bleb Appearance Grading Score (IBAGS).<sup>4,9</sup> Subjects who agree to

participate and provide written informed consent will undergo AS-OCT imaging (Spectralis OCT,

Heidelberg) of the bleb. During their operation, the Zeiss Artevo digital microscope integrated

with iOCT (Zeiss Artevo 800, Carl Zeiss Meditec AG), a commercially available device will be

utilized to visualize and evaluate the morphology of the trabeculectomy bleb at the start and

conclusion of the case.

PROCEDURES INVOLVED:

The devices used in the study are commercially available and have been used extensively in

ophthalmology and intraocular surgery. Therefore, no experimental devices will be used. The

AS-OCT is routinely obtained and is considered standard of care. The iOCT is commercially

available and is also utilized routinely in ophthalmic surgery, particularly for retinal surgery.

The Zeiss Artevo digital microscopy integrated with intraoperative OCT will be used as an

adjunct to TCNR. Published research<sup>4,6</sup> has not shown iOCT to increase risk of complications

associated with routine TCNR and we believe injury from imaging is not biologically plausible.

Surgery and iOCT will be recorded and saved to a secure NMH server. The surgical videos will

only be used for research purposes.

Review of medical records will be performed for patients who agree to participate in the

prospective study. Data gathered will include basic demographic information and clinical data

relevant to glaucoma management (visual acuity, intraocular pressure, medications, disease

Version Date: 04/16/2021

 HRP-593 / v03152019

STU00213080

severity). Post-operative course including intraocular pressure, intraoperative or post-operative

complications and repeat TCNR or additional surgery will also be collected.

Furthermore, a retrospective review of medical records will be performed for patients who

underwent TCNR without iOCT or AS-OCT assistance by the same surgeon during the period

from June 1, 2015 to June 1, 2020. This group of patients will serve as historical controls. These

individuals will be identified using Enterprise Data Warehouse and billing data. We aim to

identify approximately 25 controls. The selection criteria for controls are 1) age within 5 years

of each study patient 2) same race as study patient 3) diagnosis of open angle glaucoma and 4)

adequate follow up of at least 3 months.

**DATA AND SPECIMEN BANKING** 

Participants will be assigned a study ID. The patient identifiers will be stored separately from

the coded study data.

Data abstracted from the medical record will be collected on a secure sever, with computers

only accessible with passwords. Only the research team will have access to the identified data.

**SHARING RESULTS WITH PARTICIPANTS** 

The results are part of the standard glaucoma care for each participant and they will be

discussed with participants as part of the management of the condition.

**STUDY TIMELINES** 

Version Date: 04/16/2021

 HRP-593 / v03152019

STU00213080

The participant will be in the study for the duration of their office visit (with AS-OCT testing)

and surgery. In the context of this research study, participants will also be followed for 12

months after surgery to assess their post-operative course.

It will likely take approximately 12 months to enroll all study participants. The estimated date

for completion of primary analyses will be 6 months after enrollment of study.

**INCLUSION AND EXCLUSION CRITERIA** 

Inclusion criteria

Briefly, the diagnosis of glaucoma is based on the presence of 2 or more of the following

findings: 1) glaucomatous optic disc damage, defined as the presence of optic disc

excavation, diffuse or focal neuroretinal rim thinning or notching, localized or

generalized RNFL thinning; 2) visual field defects consistent with glaucoma; and 3) IOP ≥

22 mmHg.

Patients with glaucoma who have been advised to undergo TCNR of a failed

trabeculectomy bleb by a glaucoma specialist at Northwestern Medicine

History of failed trabeculectomy (based on clinical features of the trabeculectomy bleb)

and elevated intraocular pressure)

Patients can have history of other glaucoma surgery or cataract surgery

The diagnosis of glaucoma is based on the presence of 2 or more of the following

findings: 1) glaucomatous optic disc damage, defined as the presence of optic disc

excavation, diffuse or focal neuroretinal rim thinning or notching, localized or

generalized RNFL thinning; 2) visual field defects consistent with glaucoma; and 3) IOP ≥

22 mmHg.

Exclusion criteria

Age younger than 18 years;

Secondary causes of glaucoma (e.g., iridocyclitis, trauma);

- Any evidence of corneal or conjunctival pathology adjacent to filtration bleb that could influence AS-OCT image
- Patients who did not undergo surgery or have adequate follow up
- Adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, prisoners and vulnerable populations

## **VULNERABLE POPULATIONS: NONE**

# **PARTICIPANT POPULATION(S)**

**Prospective Study Population** 

| Accrual | Category/Group: | Consented: | Enrolled: |
|---|---|---|---|
| Number: | (Adults/Children | Maximum Number to be | Number to |
| | Special/Vulnerable | Consented or | Complete the Study |
| | Populations) | Reviewed/Collected/Screened | or Needed to |
| | | | Address the |
| | | | Research Question |
| Local | 25 adults | 25 adults | 25 eyes |
| Study-wide | | | |
| Total: | 25 adults | 25 adults | 25 eyes |

Age and race matched historical controls (identified via retrospective chart review)

| Accrual | Category/Group: | Consented: | Enrolled: |
|---|---|---|---|
| Number: | (Adults/Children | Maximum Number to be | Number to |
| | Special/Vulnerable | Consented or | Complete the Study |
| | Populations) | Reviewed/Collected/Screened | or Needed to |
| | | | Address the |
| | | | Research Question |

Version Date: 04/16/2021  HRP-593 / v03152019

| Local | 25 adults | 0 | 25 eyes |
|------------|-----------|---|---------|
| Study-wide | | | |
| Total: | 25 adults | 0 | 25 eyes |

### **RECRUITMENT METHODS**

Potential participants will be identified from the patients scheduled for follow up in the Glaucoma Service at Northwestern Medicine. Potential participants who are already scheduled for surgery may be called to gauge interest in the study. If they express interest, the patient will return to clinic prior to surgery to review and sign the informed consent and complete presurgery study imaging. Only patients who fit the inclusion/exclusion criteria will be asked to participate in the study.

## **COMPENSATION FOR PARTICIPATION IN RESEARCH ACTIVITIES**

There is no additional cost for the patient to participate in this study. Patients and their insurance companies will be billed for office visits and procedures that are part of their usual medical care. There is no compensation made to the study subjects for participating in this study. Patients will have routine preoperative and postoperative follow up visits as necessary based on their clinical course. No extra visits will be required as a result of participation in this study.

## WITHDRAWAL OF PARTICIPANTS

All the participants are free to withdraw at any point of the study. In case the participants are not willing to continue with the study protocol they will be removed from the analysis.

### **RISKS TO PARTICIPANTS**

Version Date: 04/16/2021  HRP-593 / v03152019

STU00213080

There is a risk of loss of confidentiality of the information that is used in this study. To minimize

the risk of breach in confidentiality, the consent process for the prospective study will be done

in a private room. Patient names will be replaced with arbitrary IDs. For the duration of the

study, the patients will be referred by their ID. All data will be kept in a password-protected file.

POTENTIAL BENEFITS TO PARTICIPANTS

There may be no direct benefits of this study to the patient. Results of this study may provide

important knowledge that will be generalizable to the care of other patients with glaucoma.

DATA MANAGEMENT AND CONFIDENTIALITY

PROVISIONS TO MONITOR THE DATA TO ENSURE THE SAFETY OF PARTICIPANTS

For the prospective study, the consent process and all the study procedures will be done in a

private room/space. To protect participant's confidentiality, their information and study

conduct will only be discussed with individuals listed in the study personnel.

In general, patients' data and all information pertaining to this study will remain confidential

and all the study materials will be kept in a password protected computer a password-

protected file and a secure server. Paper files will be kept in a locked drawer. In addition, the

identifier list will be maintained separately from the study data. This identifier list will be kept in

a password-protected file on a secure server.

PROVISIONS TO PROTECT THE PRIVACY INTERESTS OF PARTICIPANTS

The study is done in the same facility that glaucoma clinic is located and patients are imaged

with the AS-OCT device on the same floor. The acquired data with AS-OCT are similar to images

routinely taken for their glaucoma follow up. The iOCT is attached to the operating microscope

in the same operating room that is routinely used for ocular surgery. The consent process and

STU00213080

all the study procedures for individuals enrolled in the prospective study will be done in a

private room/space.

To protect participant's confidentiality, their information and study conduct will only be

discussed with individuals listed in the study personnel. Patients' data and all information

pertaining to this study will remain confidential and all the study materials will be kept in a

password-protected computer a password-protected file and a secure server. Paper files will be

kept in a locked drawer.

**COMPENSATION FOR RESEARCH-RELATED INJURY** 

This study is minimal risk and therefore, there will be no anticipated research related injuries in

this study or compensation for such injuries

**ECONOMIC BURDEN TO PARTICIPANTS** 

Patients will be billed for the office visit as this was planned in advance. There will be no extra

cost to patients as a result of this study. The AS-OCT or iOCT that will be performed as part of

this study will not be billed to the patient or their insurance carrier.

**CONSENT PROCESS** 

Potential participants in the prospective study will be identified from the patients scheduled for

follow up or surgery in the Glaucoma Service at Northwestern Medicine. Patients will be

approached verbally about the study during their visits or over the phone by study approved

personnel. The informed consent process will take place in person in a private room. The

research team will go over the consent forms with the patients to ensure they understand the

nature of the research study, its procedures, potential risks and benefits, and their

responsibilities as participants. The patients will be given as much time as needed to consider

the study and address any questions or concerns. If patients need additional time to decide

whether or not to enroll in the study, they will have the option of rescheduling for a later time.

Version Date: 04/16/2021

 HRP-593 / v03152019

STU00213080

Throughout the consent process, the research team will stress that participation is completely

voluntary and that participants may withdraw from the study at any point. Patients will be

provided a copy of the fully executed, signed consent forms. An additional copy of the signed

consent forms will be scanned into the patient's electronic medical record and hard copies will

be maintained in the subject binder.

For the historical control data, a retrospective chart review of glaucoma patients who

underwent TCNR surgery from June 1, 2015 to June 1, 2020, will be performed. Consent will not

be obtained for these patients as they will not undergo any further testing or treatments.

**NON-ENGLISH SPEAKING PARTICIPANTS** 

Only English-speaking patients will be included in this study

WAIVER OR ALTERATION OF CONSENT PROCESS

Written consent form will be required for all participants; except for patients in the control

arm.

Waiver of consent is requested for subjects in the control arm.

This research involves no more than minimal risk of harm to the subjects and involves no

procedure for which written consent is normally required outside the research context.

Given the retrospective nature of the data collection and de-identified reporting, the waiver

should not adversely affect the rights or welfare of the participants. Protocols are in place to

protect information and ensure minimal risk of identifiers being improperly used or disclosed.

The waiver or alteration will not adversely affect the rights and welfare of the participants

**Process to Document Consent in Writing** 

STU00213080

For the prospective study, the consent process and all the study procedures will be done in a

private room/space. To protect participant's confidentiality, their information and study

conduct will only be discussed with individuals listed in the study personnel. The process will be

documented using the department's standard consent documentation template. It may also be

noted in Epic.

Waiver of HIPAA Authorization

Use of PHI described in the protocol is necessary to the research. The research could not

practicably be conducted without access to and use of the protected health information.

Protected health information will not be reused or disclosed to any other person or entity,

except as required by law, for authorized oversight of the research project, or for other

research for which the use or disclosure of protected health information would be permitted by

the HIPAA Privacy Rule.

Given the retrospective nature of the data collection and de-identified reporting, the waiver

should not adversely affect the rights or welfare of the participants. Protocols are in place to

protect information and ensure minimal risk of identifiers being improperly used or disclosed.

There is a plan to destroy the identifiers at the earliest opportunity consistent with conduct of

the research as described in the Access Security and Management section, unless there is a

health or research justification for retaining the identifiers.

PROTECTED HEALTH INFORMATION

Participant will be assigned a study ID. The patient identifiers will be stored separately from the

coded study data.

Data abstracted from the medical record will be collected on a secure sever, with computers

only accessible with passwords. Only the research team will have access to the identified data

**ACCESS SECURITY AND MANAGEMENT** 

Subjects will be assigned a coded number and a coded identifier list with the corresponding

name to an identification number will be kept in locked files in the ophthalmology department,

STU00213080

of which only authorized research personnel will have access to. The data recorded for the

study will be kept as a password-protected file on a password protected computer, separate

from the subject log key. Data will be recorded and analyzed in a coded manner, with only

authorized research personnel having access to it. Health information collected during the

study will be stored electronically in password-protected files in the Department of

Ophthalmology and then will be deleted at the earliest opportunity at the close of the study

and no later than 10 years.

QUALIFICATIONS TO CONDUCT RESEARCH AND RESOURCES AVAILABLE

We estimate that there are a few patients in each glaucoma clinic that qualify to be included in

the prospective study. Patients are selected among the patients that are being followed for

glaucoma in the glaucoma clinic. The clinical examination is done as part of the routine

glaucoma follow up and imaging will be acquired at the same day. Imaging with devices will

take few minutes and do not pose any risk to patients.

The eye clinic at Northwestern University has qualified and trained staff. Dr. Angelo Tanna is a

Professor and Vice Chairman in the Department of Ophthalmology at Northwestern University

and has 20 years of experience in Ophthalmology practice. He, along with his team of

ophthalmologist colleagues and fellows will recruit, verbally consent, collect anonymous

responses and analyze data.

In addition, Dr. Angelo Tanna and the other co investigators will ensure the proper adherence

to this protocol and data reviewing. All IRB approved staff involved with the study will be given

access to the protocol and trained on their roles/responsibilities.

REFERENCES

1. Arora KS, Robin AL, Corcoran KJ, Corcoran SL, Ramulu PY. Use of Various Glaucoma Surgeries and Procedures in Medicare Beneficiaries from 1994 to 2012. *Ophthalmology*.

2015;122(8):1615-1624.

2010)122(0).1010 102 ...

2. Kirwan JF, Lockwood AJ, Shah P, et al. Trabeculectomy in the 21st century: a multicenter

analysis. Ophthalmology. 2013;120(12):2532-2539.

Version Date: 04/16/2021 

HRP-593 / v03152019

- 3. Mastropasqua R, Fasanella V, Agnifili L, Curcio C, Ciancaglini M, Mastropasqua L. Anterior segment optical coherence tomography imaging of conjunctival filtering blebs after glaucoma surgery. *BioMed research international*. 2014;2014:610623.
- 4. Hamanaka T, Omata T, Sekimoto S, Sugiyama T, Fujikoshi Y. Bleb analysis by using anterior segment optical coherence tomography in two different methods of trabeculectomy. *Investigative ophthalmology & visual science.* 2013;54(10):6536-6541.
- 5. Kojima S, Inoue T, Kawaji T, Tanihara H. Filtration bleb revision guided by 3-dimensional anterior segment optical coherence tomography. *Journal of glaucoma*. 2014;23(5):312-315.
- 6. Ehlers JP, Modi YS, Pecen PE, et al. The DISCOVER Study 3-Year Results: Feasibility and Usefulness of Microscope-Integrated Intraoperative OCT during Ophthalmic Surgery. *Ophthalmology.* 2018;125(7):1014-1027.
- 7. Dada T, Angmo D, Midha N, Sidhu T. Intraoperative Optical Coherence Tomography Guided Bleb Needling. *Journal of ophthalmic & vision research.* 2016;11(4):452-454.
- 8. Kumar RS, Jariwala MU, V SA, et al. A Pilot Study on Feasibility and Effectiveness of Intraoperative Spectral-Domain Optical Coherence Tomography in Glaucoma Procedures. *Translational vision science & technology.* 2015;4(2):2.
- 9. Cantor LB, Mantravadi A, WuDunn D, Swamynathan K, Cortes A. Morphologic classification of filtering blebs after glaucoma filtration surgery: the Indiana Bleb Appearance Grading Scale. *Journal of glaucoma*. 2003;12(3):266-271.

Version Date: 04/16/2021  HRP-593 / v03152019